CLINICAL TRIAL: NCT02206126
Title: Effects of Energy Restriction on Sleep Apnea, Sympathetic Activity, Oxidative Stress, Inflammatory Biomarkers, Endothelial Function, Body Adiposity, Metabolic Profile and Blood Pressure in Obese Patients With Obstructive Sleep Apnea
Brief Title: Weight Loss and Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Antonio Felipe Sanjuliani, Antonio Felipe Sanjuliani, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLINEX05
Record Dates: First submitted 2014-06-27; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Weight loss; Obesity; Sympathetic activity; Metabolic profile; Endothelial function
MeSH Terms: conditions — Sleep Apnea, Obstructive; Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Energy restriction group (Experimental): The energy restriction group was instructed to follow an energy-restricted diet (-800 kcal/day).
  Interventions: Behavioral: Energy Restriction
- Control group (No Intervention): The control group was advised not to change their food intake.

INTERVENTIONS:
Behavioral: Energy Restriction — The energy restriction group was instructed to follow an energy-restricted diet (-800 kcal/day).
  Arms: Energy restriction group

SUMMARY:
The purpose of this study is to evaluate the effects of moderate energy restriction on the body adiposity, severity of OSA, blood pressure, sympathetic activity, oxidative stress, inflammatory biomarkers, metabolic profile and endothelial function in obese patients with OSA.

DETAILED DESCRIPTION:
Introduction: Nutritional intervention for weight loss is one of the treatment options for obstructive sleep apnea (OSA) in patients with excess body adiposity. However, the effects of moderate energy restriction, recommended by current guidelines for the treatment of obesity, on OSA are not yet known. Objective: To evaluate the effects of moderate energy restriction on the body adiposity; severity of OSA; blood pressure; sympathetic activity; oxidative stress; inflammatory biomarkers; metabolic profile and endothelial function in obese patients with OSA. Methods: A 16-week randomized clinical trial, involving 21 subjects with obesity (grade I or II), aged 20-55 years and presenting an apnea/hipopnea index (AHI) > 5 events/h. Participants were randomized into 2 groups: 11 in the energy restriction group (ERG) and 10 in the control group (CG). The ERG was instructed to follow an energy-restricted diet (-800 kcal/day) and the CG was advised not to change their food intake. At the beginning and at the end of the study, participants underwent evaluation of: OSA with the equipment Watch- PAT200® including the determination of the following parameters of OSA severity: AHI, minimum O2 saturation, number of O2 desaturations >4%; body adiposity (weight, %body fat and circumferences of waist, hip and neck); blood pressure (BP); sympathetic nervous system activity (plasma levels of catecholamines); inflammatory biomarkers (c-reactive protein and adiponectin); oxidative stress (malondialdehyde); metabolism of glucose (glucose, insulin and HOMA-IR) and lipids (total cholesterol and fractions and triglycerides); and endothelial function (index of reactive hyperemia evaluated by Endo - PAT 2000® and cellular adhesion molecules). The statistical analysis was performed with the software STATA v. 10. The level of statistical significance was p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-55 years
* body mass index (BMI) ≥ 30 kg/m2 and < 40 kg/m2

Exclusion Criteria:

* smoking
* Use of dietary supplements
* Use of medications that could interfere in body weight, metabolic profile and blood pressure
* Use of permanent pacemaker; use of α-adrenergic blocking agents
* Recent changes (within previous 6 months) in body weight (> 3 kg), in dietary intake and in intensity or frequency of physical exercise
* Diagnosis of diabetes mellitus, hypertension, dyslipidemia (with drug treatment) and kidney disease
* Clinical history of thyroid dysfunction, angina pectoris, peripheral vascular disease, peripheral neuropathy, heart failure, liver failure, chronic pulmonary disease, gastroesophageal reflux disease, myocardial infarction and stroke; finger deformity that prevents the proper use of the sensors that are necessary to evaluate OSA and endothelial function; and previous bilateral cervical-thoracic sympathectomy
* Pregnant or lactating women were not allowed into the study

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Apnea/hipopnea index | 16 weeks

SECONDARY OUTCOMES:
Blood pressure | 16 weeks
Sympathetic activity | 16 weeks
  Plasma levels of catecholamines
Oxidative stress | 16 weeks
  Serum levels of malondialdehyde
Inflammatory biomarkers | 16 weeks
  Circulating levels of high-sensitivity C reactive protein and adiponectin
Metabolic profile | 16 weeks
  Fasting plasma glucose, insulin, total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides
Endothelial function | 16 weeks
  Circulating levels of cellular adhesion molecules (intercellular adhesion molecule 1 and P-selectin).
  Endothelial function was also evaluated by the PAT method, using Endo-PAT 2000®.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Felipe Sanjuliani, Dr., Principal Investigator — Rio de Janeiro State University
Locations (1):
- Discipline of Clinical and Experimental Pathophysiology, CLINEX, Rio de Janeiro, Rio de Janeiro, Brazil